CLINICAL TRIAL: NCT05430308
Title: A Randomized Controlled Study to Compare Chlorhexidine-Alcohol Versus Povidone-iodine for Surgical Site Preparation in Subjects Undergoing Medical Thoracoscopy for the Prevention of Infectious Complications
Brief Title: Surgical Site Preparation in Subjects Undergoing Medical Thoracoscopy
Acronym: CAPTAIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Inderpaul singh, Assistant Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INT/IEC/2018/000151
Record Dates: First submitted 2022-06-18; First posted 2022-06-24 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Medical Thoracoscopy
Keywords: thoracoscopy; surgical site infection; pleuroscopy; thoracentesis
MeSH Terms: conditions — Surgical Wound Infection | interventions — Povidone-Iodine

STUDY DESIGN:
Intervention Model Description: Open labelled parallel study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chlorhexidine-alcohol scrub (Experimental): The surgical site selected for performing the thoracoscopy will be cleaned with 4%w/v chlorhexidine gluconate solution for 3 minutes. This will then be washed with normal saline and a sterile gauge. After drying chlorhexidine gluconate (2.5%v/v)-ethanol IP (70%v/v) will be applied and allowed to dry for 3 minutes before the incision.
  Interventions: Procedure: Chlorhexidine scrub
- Povidone-iodine (Active Comparator): The surgical site selected for performing the thoracoscopy will be just cleaned with normal saline followed by 10% w/v povidone-iodine solution and would be allowed to dry for 3 minutes before the incision
  Interventions: Procedure: Povidone-iodine

INTERVENTIONS:
Procedure: Chlorhexidine scrub — Surgical site selected for performing the thoracoscopy will be cleaned with 4%w/v chlorhexidine gluconate solution for 3 minutes
  Arms: Chlorhexidine-alcohol scrub
Procedure: Povidone-iodine — The surgical site selected for performing the thoracoscopy will be just cleaned with normal saline followed by 10% w/v povidone-iodine solution
  Arms: Povidone-iodine

SUMMARY:
Medical thoracoscopy is the preferred procedure for performing pleural biopsy in patients with pleural effusions that remain undiagnosed after pleural fluid analysis. Surgical site infections (SSI) and empyema are among the important complications of the procedure.

At author's center, povidone-iodine is used for surgical site preparation during MT. The investigators hypothesized that chlorhexidine-alcohol would be superior to povidone-iodine in reducing the rate of infectious complications following thoracoscopy. In this study, the authors propose to investigate the efficacy of chlorhexidine-alcohol scrub in preventing post procedural infectious complications in subjects undergoing medical thoracoscopy

DETAILED DESCRIPTION:
Medical thoracoscopy is the preferred procedure for performing pleural biopsy in patients with pleural effusions that remain undiagnosed after pleural fluid analysis. Unlike video-assisted thoracoscopic surgery that is performed under general anesthesia and single lung ventilation, medical thoracoscopy is performed under conscious sedation and local anesthesia. Medical thoracoscopy is generally a safe procedure, albeit with a small risk of complications. Surgical site infections (SSI) and empyema are among the important complications of the procedure. Author's center is a tertiary care referral hospital; the majority of the patients are referred to the authors' center late in the course of their illness. In fact, most patients have had several thoracenteses, and many patients have pleural adhesions. The authors have observed a significant incidence of post procedural infections (7.8-10%) in previous studies. In a recent RCT, investigators have demonstrated that the prophylactic use of antibiotics did not reduce the incidence of SSI. Since the patient's skin is a major source of pathogens, it is conceivable that improving skin antisepsis would decrease surgical-site infections. The aim of preoperative skin preparation is to reduce the risk of SSIs by removing soil and transient organisms from skin. Antiseptics have the ability to bind to the skin's stratum corneum that results in persistent chemical activity on the skin. A SSI occurs when the number of bacteria at the incision site overcome the hosts immune defense mechanism. The Centers for Disease Control and Prevention (CDC) recommends that 2% chlorhexidine-based preparations be used to cleanse the site of insertion of vascular catheters. However, the CDC has not issued a recommendation as to which antiseptics should be used preoperatively to prevent postoperative SSIs.

In a previous RCT comparing preoperative cleansing of the patient's skin, chlorhexidine-alcohol was found to be superior to cleansing with povidone-iodine for preventing surgical-site infection after clean contaminated surgery. However, in a pooled analysis of 13 RCTs comparing surgical site preparation for clean surgeries, no clear benefit could be demonstrated of either agent for preventing SSIs. Also, no published randomized studies have examined the effect of one antiseptic preparation over another on the incidence of surgical-site infection during medical thoracoscopy. A recent guideline on medical thoracoscopy has no mention about the preferred agent for skin preparation during MT. At the author's center, povidone-iodine is used for surgical site preparation during MT. The authors hypothesized that chlorhexidine-alcohol would be superior to povidone-iodine in reducing the rate of infectious complications following thoracoscopy. In this study, the investigators propose to investigate the efficacy of chlorhexidine-alcohol scrub in preventing post procedural infectious complications in subjects undergoing medical thoracoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥12 <80 years
2. Medical thoracoscopy being performed for the workup of undiagnosed pleural effusion

Exclusion Criteria:

1. Patients with intercostal tube before MT
2. MT performed for adhesiolysis
3. Age <12 or ≥80 years
4. SPO2 <92% at room air
5. Hemodynamic instability
6. Myocardial infarction or unstable angina in the last 3 months
7. Hemoglobin <8g/dl; Platelet count <50,000 cell/dl
8. Lack of pleural space due to adhesions
9. Uncorrected coagulopathy (PT > 3 seconds above control; APTT> 10 seconds above control)
10. Failure to provide informed consent
11. Patients already taking any antibiotic due to any reason

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-04-18 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of infection | 30 days
  surgical site indicated by development of a purulent discharge from the incision site or pleural space infection as indicated by development of purulent fluid, fall in glucose levels or Gram stain or culture positivity in the pleural fluid drained by the chest tube on the side of the procedure

SECONDARY OUTCOMES:
Rate of adverse effects | 6 hours
  Adverse effects arising as a result of the use of either chlorhexidine-gluconate or povidone-iodine such as skin erythema, and rash
Duration of chest tube drainage | 30 days
  Time from insertion of chest tube to removal of chest tube

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - Bronchoscopy suite, PGIMER, Chandigarh
  - Bronchoscopy suite, Chandigarh

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared on request to the PI